CLINICAL TRIAL: NCT05905510
Title: Comparative Study Between Ultrasound-Guided Lumbar Erector Spinae Plane Block and Fascia Iliaca Compartment Block for Postoperative Analgesia After Total Hip Arthroplasty
Brief Title: Lumbar Erector Spinae Plane Block and Fascia Iliaca Compartment Block After Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ahmed Zahran, Doctor Ahmed Ahmed Eldemrdash Zahran Resident of Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine,Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35153/12/21
Record Dates: First submitted 2023-05-18; First posted 2023-06-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (Active Comparator): Patients will receive spinal anesthesia alone (30 ml bupivacaine 0. 25%).
  Interventions: Drug: spinal anesthesia plane block
- Lumbar Erector spinae plane block (L-ESPB) (Active Comparator): Patients will receive spinal anesthesia and then ipsilateral lumbar erector spinae plane block (30 ml bupivacaine 0. 25%) at the level of the lumbar region in the operating room after the end of the surgery.
  Interventions: Drug: Lumbar Erector spinae plane block (L-ESPB)
- Fascia iliaca compartment block (FICB) (Active Comparator): Patients will receive spinal anesthesia and then ipsilateral suprainguinal fascia iliaca compartment block (30 ml bupivacaine 0. 25%) in the operating room after the end of the surgery.
  Interventions: Drug: Fascia iliaca compartment block (FICB)

INTERVENTIONS:
Drug: Lumbar Erector spinae plane block (L-ESPB) — The fourth lumbar vertebral level will be determined using the conventional method (the imaginary line between two crista iliacas). The convex transducer will be placed at the mid-vertebral line in the sagittal plane. The transducer will be shifted from the midline, 3.5-4 cm laterally, to the side of the surgery to visualize the erector spinae muscle and transverse process. Using the out-of-plane technique, a 22G/80-mm block needle will be advanced until it reached the transverse process. 0.5-1 ml of the prepared local anesthesia solution (30 ml bupivacaine 0.25%) will be administered, leading to hydro dissection to confirm the correct location. The needle will be repositioned by pulling back a few millimeters if resistance occurred when administering local anesthesia. All local anesthesia will be administered to this location between the transverse process and the erector spinae muscle
  Arms: Lumbar Erector spinae plane block (L-ESPB)
Drug: Fascia iliaca compartment block (FICB) — The transducer will be placed laterally to the femoral nerve. It then rotated 90 degrees to the sagittal plane, under ultrasound guidance, a regional block needle (22 G, 80 mm) will be introduced in the cranial direction. Once good needle alignment with the ultrasound beam is achieved, the needle will be inserted deep into the tissues until an optimal position of the needle tip is obtained. Needle location will be additionally verified by injecting 0.5-1 ml of the prepared local anesthesia solution and observing the solution spread within the tissues. Once the correct position of the needle tip is confirmed, the local anesthetic will be deposited under the iliac fascia to force its flow towards the lumbar plexus. 30 ml of bupivacaine 0.25% solution will be used for the block. local anesthesia will be administered as 5 mL boluses with a 20 second interval.
  Arms: Fascia iliaca compartment block (FICB)
Drug: spinal anesthesia plane block — Patients will receive spinal anesthesia alone
  Arms: Control Group

SUMMARY:
Compare the analgesic efficacy of ultrasound-guided lumbar erector spinae plane block (L-ESPB) versus fascia iliaca compartment block (FICB) in patients scheduled for total hip arthroplasty.

DETAILED DESCRIPTION:
Ultrasound-guided erector spinae plane (ESP) block is a recent regional anesthetic technique. It was first described by Forero et al. in 2016 for acute and chronic thoracic pain management. Local anesthetic (LA) is injected between the erector spinae muscle and the vertebra's transverse process, leading to the spread of LA cephalad, caudally, and through the paravertebral space.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 30-75 years from both sexes.
2. ASA I-III scheduled for unilateral hip surgery under spinal anesthesia.

Exclusion Criteria:

1. Patients' refusal.
2. Patients who were unable to co-operate with researchers.
3. History of allergy to local anesthetics.
4. Local infection at the site of the block.
5. Patients with bleeding and coagulation disorders.
6. Patients with renal, hepatic, cardiac decompensation, or spine deformities.
7. Patients receiving opioids for chronic analgesic therapy
8. Body mass index > 35 kg/m2

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative pain | UP to 24 hour postoperatively
  Assessment of postoperative pain using the Numeric rating scale (NRS), NRS is a valid and simple approach to pain assessment (0= no pain and 10= worst possible pain)

SECONDARY OUTCOMES:
Time required for the first rescue analgesia. | Up to 24 hours postoperatively
  Morphine sulfate 0.03 mg/kg will be administered intravenous as a rescue analgesic if Numeric rating scale is ≥ 4
The total postoperative rescue analgesic | first 24 hours postoperatively
  The total amount of morphine consumption
Adverse effects | Up to 24 hours postoperatively
  Any complications or undesirable side effects will be observed and treated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author from one year after study completion
Supporting Information: Study Protocol
Time Frame: From one year after study completion
Access Criteria: The data will be available upon reasonable request from the corresponding author.